CLINICAL TRIAL: NCT01604681
Title: The Effect of Flaxseed Oil Supplementation on Biomarkers, Quality of Life and Cognitive Function in Hypertensive and Dyslipidemic Subjects With or Without the C677T and A1298C Polymorphisms in MTHFR Gene in Different Municipalities of Rio de Janeiro
Brief Title: Supplementation With Flaxseed Oil in the State of Rio de Janeiro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ana Paula Alves Avelino, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 171/2011
Record Dates: First submitted 2012-05-18; First posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension; Dyslipidemia
Keywords: Linseed Oil; Oxidative Stress; Polymorphism, Genetic; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Dyslipidemias; Cardiovascular Diseases | interventions — Control Groups; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator): 3 g of powdered gelatin encapsulated in opaque capsules.
  Interventions: Dietary Supplement: Placebo
- Flaxseed oil group (Experimental): Oil extracted from linseed by pressing the cold and encapsulated, providing 3g per day containing 1.75 g of alpha linolenic acid.
  Interventions: Dietary Supplement: Flaxseed Oil

INTERVENTIONS:
Dietary Supplement: Placebo — 6 capsules per day, thirty minutes before lunch and dinner, eating 3 capsules (3 g) at a time.
  Other Names: Control group
  Arms: placebo group
Dietary Supplement: Flaxseed Oil — 6 capsules per day, thirty minutes before lunch and dinner, eating 3 capsules (3 g) at a time.
  Other Names: Linseed Oil
  Arms: Flaxseed oil group

SUMMARY:
The purpose of this study is to evaluate the effect of supplementation with flaxseed oil combined with a nutritional counseling in reducing cardiovascular risk factors in homocysteine , biomarkers of inflammation, oxidative stress, improving quality of life and cognitive decline in hypertensive and dyslipidemic genotyped for the C677T and A1298C polymorphisms of methylenetetrahydrofolate reductase gene.

DETAILED DESCRIPTION:
Epidemiological data show that there is a decline in death from cardiovascular disease (CVD) in the state of Rio de Janeiro, but this did not happen in the cities of Itaperuna, Niterói and Volta Redonda, in spite of presenting different epidemiological characteristics, still have high rates of death CVD. What led to our interest in investigating these municipalities. Our goal is to evaluate the effect of supplementation with flaxseed oil combined with nutritional counseling in reducing cardiovascular risk factors in homocysteine, biomarkers of inflammation, oxidative stress, improving quality of life and cognitive decline in hypertensive individuals dyslipidemic and genotyped for polymorphisms C677T and A1298C methylenetetrahydrofolate reductase gene (MTFHR). This is a clinical trial, double blind, placebo-controlled, randomized block, lasting three months. Study participants will be recruited from August 2011 to August 2013. Will be recruited at least 200 individuals in each city, considering possible losses and ensuring consistent results. Subjects will be randomized in blocks of 10, five patients in the group supplemented with linseed oil and five patients in the control group with placebo supplementation, ensuring proper distribution of the number of participants in the study groups. Will be collecting information on the socio-economic status of study participants through a structured questionnaire will be carried out assessment of food consumption - frequency of consumption and 24 hours, clinic - blood pressure, anthropometric - height, weight, waist circumference and BMI, body composition - bioelectrical impedance analysis, biochemical tests - lipid profile, blood glucose, insulin, homocysteine, serum folate concentrations in erythrocytes and, cobalamin, vitamin C, E and A, minerals - zinc, iron, copper and selenium, markers of oxidative stress and inflammatory response and molecular analysis - C677T and A1298C polymorphisms of methylenetetrahydrofolate reductase gene. It will also be diagnosed with depression and evaluation of physical activity and quality of life using questionnaires were previously validated. Our results demonstrate the effectiveness of supplementation with flaxseed oil, in reinforcing the results of nutritional counseling in reducing cardiovascular risk factors and biomarkers studied, besides adding to the knowledge about the interactions between markers of inflammation, oxidative stress with oil supplementation flaxseed and polymorphisms C677T and A1298C MTHFR gene, on which there are no reports in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension and/or dyslipidemia,
* Have over 20 years,
* Both sexes,
* Any skin color and
* Take part in the study by signing the consent form.

Exclusion Criteria:

* Make use of some food or vitamin supplement,
* HIV positive and cancer.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Polymorphisms | Up to 3 months
  To evaluate the effect of nutritional counseling associated with linseed oil supplementation on biomarkers estutados according to the C677T and A1298C polymorphisms of the MTHFR gene.

SECONDARY OUTCOMES:
Cognitive decline | Up to 3 months
  To evaluate the effect of nutritional counseling associated with linseed oil supplementation on cognitive decline.
Quality of life | Up to 3 months
  To evaluate the effect of nutritional counseling associated with linseed oil supplementation on Quality of life.
Oxidative stress | Up to 3 months
  To evaluate the effect of nutritional counseling associated with linseed oil supplementation on biomarkers of oxidative stress.
Lipid profile | Up to 3 months
  To investigate the effect of supplementation of flaxseed oil combined with nutritional guidance on lipid profile, according to the consumption of saturated fat.

CONTACTS AND LOCATIONS:
Locations (1):
- Clementino Fraga Filho University Hospital Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil